CLINICAL TRIAL: NCT04246268
Title: Assessment of the INVOcell Intravaginal Culture System During 5-day (120 Hours) Vaginal Incubation
Brief Title: Assessment of the INVOcell Intravaginal Culture System
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: INVO Bioscience is suspending trial per ASRM's recommendations during Covid-19 pandemic.
Sponsor: INVO Bioscience, Inc. (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-017
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Device: INVOcell Intravaginal Culture System
  Intervention: During an IVF/IVC cycle, participants will retain the INVOcell Culture Device with the Retention Device in the vaginal cavity for 5-days vaginal incubation.
  Interventions: Device: INVOcell

INTERVENTIONS:
Device: INVOcell — Female participants undergoing in vitro fertilization (IVF) and/or Intracytoplasmic Sperm Injection (ICSI) for assisted reproduction will be asked to participate.
  Other Names: Intravaginal Culture; IVC; Vaginal Incubation

SUMMARY:
The INVOcell intravaginal culture system is a prescription device intended for preparing, holding, and transferring human gametes or embryos during intravaginal in vitro fertilization or intravaginal culture procedures.

The original (FG-002) INVOcell culture system was FDA cleared through De Novo application (DEN150008). The purpose of this study is to evaluate the INVO Bioscience modified INVOcell system, comprised of the INVOcell Intravaginal Culture Device and Retention Device, in terms of the following:

2.1 Effectiveness of achieving fertilization, implantation, embryo development, clinical pregnancy, and live birth after 5-days of continuous vaginal incubation.

2.2 The comfort and retention of the INVOcell device and retention system intravaginally.

DETAILED DESCRIPTION:
This is a Pivotal, single arm, multicenter, open label trial to evaluate the efficacy, comfort and retention of the INVOcell Intravaginal Culture Device and Retention Device over 5-days vaginal incubation. The effectiveness of the INVOcell device will be tested on a select population of infertile couples at several in vitro fertilization (IVF) centers. The providers at each center will conduct the processes of ovarian stimulation, egg retrieval and embryo transfer per the standard protocols for their centers. The planned sample size is 180 participants across 3 sites (60 participants per site).

The objective of this study is to assess the efficacy, comfort and retention of the INVOcell with the retention device, and demonstrate superiority following 5-day vaginal incubation as compared to current 3-day vaginal incubation indication.

Specifically, the following will be assessed:

1. The INVO Procedure using the INVOcell Intravaginal Culture Device can effectively maintain 5-days of continuous vaginal incubation with the transfer of blastocyst(s) at the end of the 5-days.
2. The Retention Device retains the INVOcell in the vaginal cavity and is well tolerated during the 5-days of continuous vaginal incubation.

ELIGIBILITY:
Inclusion Criteria:

Women diagnosed with:

* Tubal factor
* Endometriosis (stage I or II)
* Ovulatory dysfunction
* Multiple female factors
* Males with mild male factor [mild male factor is defined as meaning: two or more semen analyses that have one or more variables which fall below the 5th centile as defined by the World Health Organization (WHO, 2010)]

Couples with:

* Unexplained Infertility
* Multiple factors, of female and/or male origin

The pre-selected couples will be included in the study only if they fulfill the more specific inclusion and exclusion criteria below:

* Couples may be included in the study only if they have been informed about the study and have given their written consent.
* Infertile couples with failure to conceive a diagnosed pregnancy after one year of unprotected intercourse (6 months if the woman's age is 35 years or more). This one-year requirement need not be fulfilled if oligomenorrhea or tubal factor is present, or donor sperm use is planned
* IVF has been determined by the physician to be their next appropriate treatment
* Women with desire for pregnancy using donor sperm will be eligible even absent infertility factors.

Women included in the study should:

* Be between the age of 18 and 37 years (has not reached her 38th birthday at the time of enrollment).
* Have an anti-Müllerian hormone (AMH) level ≥ 0.8 ng/mL
* Have a normal uterine cavity as assessed in the past year by HSG, SHG or hysteroscopy. Prior tubal ligation is acceptable.
* Partner semen analysis within the past year must show a total of ≥ 15 million motile spermatozoa.

Exclusion Criteria:

* Inability to read and speak English fluently
* One (1) or more recurrent vaginitis or bacterial vaginosis (BV) requiring medical attention.
* A history of toxic shock syndrome
* Known allergies to plastic or silicone
* Had pelvic surgery within the past 8 weeks, excluding laparoscopy with or without salpingectomy (ies) or hysteroscopy with or without polypectomy
* Had pelvic inflammatory disease (PID) within the past 3 months and were treated with antibiotics
* Severe endometriosis (stage III-IV) or endometrioma(s) (past or present)
* Clinical signs of current vaginal infection
* Significant abnormalities of the vaginal cavity
* Submucous or intramural fibroids (>2 cm diameter)
* Hydrosalpinx
* Uncontrolled chronic illness, e.g. autoimmune disease, diabetes. Appropriately treated hypothyroidism, hypertension, dyslipidemia, e.g., are not exclusions.
* BMI >36.0 kg/m2
* Donor oocytes
* Antral follicle count (AFC; at cycle baseline) < 6
* Previously assessed as having a poor response to ovarian stimulation
* Patients with polycystic ovary syndrome (PCOS) meeting NIH (1990) criteria
* Cervical stenosis
* Recurrent pregnancy loss defined by recurrent non-biochemical pregnancy losses
* Failed fertilization of all oocytes obtained in a previous IVF cycle
* Smoke tobacco or vape, abuse drugs or alcohol
* Inability to understand or comply with trial procedures
* Partner with vasectomy reversal
* Partner with inability to produce sperm specimen
* Partner with uro-genital infection

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | at 7 weeks of gestation
  Clinical pregnancy rate: number of clinical pregnancies at 7 weeks of gestation divided by the number of successful egg retrieval procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Doody, MD, Study Director — INVO Bioscience, Inc.
Locations (4):
- United States (4):
  - Piedmont Reproductive Endocrinology Group, Greenville, South Carolina
  - Piedmont Reproductive Endocrinology Group, West Columbia, South Carolina
  - Fertility Center of San Antonio, San Antonio, Texas
  - The New Hope Center for Reproductive Medicine, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.